CLINICAL TRIAL: NCT05992779
Title: RELEVANCE OF COCHLEAR IMPLANTATION IN THE VERY ELDERLY: LENGTH OF DURATION AND OUTCOMES
Brief Title: Cochlear Implantation in the Elderly
Acronym: RCIVELDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0758
Record Dates: First submitted 2023-07-26; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Cochlear; Implant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient elderly implanted: Patients over 80 years old, primo implanted between 2011 and 2021
  Interventions: Other: Measuring the vocal audiometry of patients.; Other: Measuring data loging

INTERVENTIONS:
Other: Measuring the vocal audiometry of patients. — Measuring vocal audiometry at 6 months, 1 year and annually until the last date of follow-up
Other: Measuring data loging — Measuring data loging at 6 months, 1 year and then annually until last date of follow-up

SUMMARY:
The goal of this study is to demonstrate that cochlear implantation is an effective, reasonable, and viable long-term option within a very elderly population

ELIGIBILITY:
* Inclusion Criteria :

  * 80 years or more
  * Primo-implantation
* Exclusion Criteria :

  * Under 80 years
  * Bilateralisation
  * Explantation or re-implantation

Min Age: 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients 80 years or more
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Vocal audiometry | Through study completion, an average of 1 year
Data Loging | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France